CLINICAL TRIAL: NCT03464981
Title: Observational Hemodynamic Monitoring During LVAD Implantation Among
Brief Title: Observational Hemodynamic Monitoring During LVAD Implantation Among Individuals With Advanced Heart Failure
Acronym: BATMAN
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 17-2119
Record Dates: First submitted 2018-02-05; First posted 2018-03-14 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Heart Failure; Circulatory Disorders Postprocedural Complication; Cardiomyopathy, Congestive; Surgery
MeSH Terms: conditions — Heart Failure; Cardiomyopathy, Dilated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Advanced HF patients scheduled to undergo LVAD implantation

SUMMARY:
The overall objective of this pilot analysis is to characterize the hemodynamic changes that occur during implantation of a left ventricular assist device (LVAD) in patients with advanced heart failure - specifically, how right ventricular function is compromised as a result of LVAD implantation.

ELIGIBILITY:
Inclusion Criteria:

* individuals ≥ 18 years of age with severe heart failure (HF) and who have been approved by the advanced HF selection committee for LVAD implantation.

Exclusion Criteria:

* Patients with pre-existing right ventricular (RV) dysfunction/failure, defined as:

  1. Imaging evidence of moderate-severe RV dysfunction on echocardiography
  2. Hemodynamic evidence of RV dysfunction with:

     * a right-atrial pressure (RAP): pulmonary capillary wedge pressure (PCWP) ratio of ≥ 0.67 (note: this index compares pressures on the right [RAP] and left [PCWP] side of the heart;
     * an RAP/PCWP ratio ≥ 0.67 provides hemodynamic evidence of RV dysfunction.
  3. Clinical evidence of preexisting RV dysfunction, as indicated by significant (3-4+ peripheral edema) and/or elevated jugular venous pressures on clinical examination.
  4. Patients with end-stage renal disease requiring hemodialysis
  5. Patients requiring temporary hemodynamic support prior to LVAD implantation with temporary LVADs, and/or veno-arterial extracorporeal membrane oxygenators ("ECMO").
  6. Planned concurrent implantation of right ventricular assist device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced HF who are scheduled to undergo LVAD implantation with either the Heartmate 2, Heartmate 3 (Abbott, Abbott Park, IL) or HVAD (Medtronic, Minneapolis, MD) LVADs
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Cardiovascular hemodynamics (invasive and noninvasive) | During LVAD implant and for 12-24 hours during ICU admission
  Cardiovascular hemodynamics will be measured both invasively and noninvasively as standard-of-care during LVAD implantation in the Operating Room (OR), and immediately afterwards in the CT-ICU unit prior to discharge.
Change in Heart Rate (HR) | During LVAD implant and for 12-24 hours during ICU admission
  Changes in HR will be evaluated during LVAD implantation in the OR, and immediately afterwards in the CT-ICU unit prior to discharge.
Change in Blood Pressure (BP) | During LVAD implant and for 12-24 hours during ICU admission
  Changes in BP will be evaluated during LVAD implantation in the OR, and immediately afterwards in the CT-ICU unit prior to discharge.
Change in Right Atrial (RA) pressure | During LVAD implant and for 12-24 hours during ICU admission
  Changes in RA pressure will be evaluated during LVAD implantation in the OR, and immediately afterwards in the CT-ICU unit prior to discharge.
Change in pulmonary pressure | During LVAD implant and for 12-24 hours during ICU admission
  Pulmonary pressure changes will be evaluated during LVAD implantation in the OR, and immediately afterwards in the CT-ICU unit prior to discharge.
Change in Cardiac output | During LVAD implant and for 12-24 hours during ICU admission
  Cardiac output changes will be evaluated during LVAD implantation in the OR, and immediately afterwards in the CT-ICU unit prior to discharge.

SECONDARY OUTCOMES:
Change in Right ventricular function | During LVAD implant and for 12-24 hours during ICU admission
  Right ventricular function will be evaluated during LVAD implantation in the OR, and immediately afterwards in the CT-ICU unit prior to discharge.
Change in Brain blood flow | During LVAD implant and for 12-24 hours during ICU admission
  Brain blood flow will be evaluated during LVAD implantation in the OR, and immediately afterwards in the CT-ICU unit prior to discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Jay D Pal, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No